CLINICAL TRIAL: NCT07000942
Title: Diagnostic Electrical Cardioversion for Explaining Patient's AF and HF Symptoms
Acronym: DEEP-AF-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M. Rienstra (Other)
Collaborators: Martini Hospital Groningen (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor-Investigator, M. Rienstra, Prof. Dr., University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DEEP-AF-HF
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF); Heart Failure (HF); Electrical Cardioversion
Keywords: Electrical cardioversion; Quality of Life (QoL); Treatment changes
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Electric Countershock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: We will use independent blinded endpoint committee to evaluate treatment changes by the physician in both treatment groups. We will provide a primary endpoint charter for the blinded endpoint committee, in which the treatment changes will be specified. Also, an adjudication committee will assess the ECGs at 4 weeks to assess the secondary endpoint; recurrences of AF.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical cardioversion (ECV) (Active Comparator)
  Interventions: Other: Electrical cardioversion (ECV)
- Standard of Care (SoC) (No Intervention)

INTERVENTIONS:
Other: Electrical cardioversion (ECV) — Electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure
  Arms: Electrical cardioversion (ECV)

SUMMARY:
Rationale:

The co-existence of Atrial Fibrillation (AF) and Heart Failure (HF) is associated with increased morbidity, mortality, and hospital admissions, significantly contributing to healthcare burden. Patients often experience overlapping symptoms, complicating identifying the disease primarily responsible for symptom burden. Electrical cardioversion (ECV) has been suggested to assess symptom status in sinus rhythm. However, the role of a diagnostic ECV in patients with AF and concomitant HF has not been established.

The hypothesis of this trial is that a diagnostic ECV can provide insight into AF-specific and HF-specific symptoms that can inform the physician and subsequently lead to treatment changes, as well as improve quality of life (QoL), and result changes in ejection fraction, cardiac output, and NT-proBNP levels.

Objective: To assess whether a diagnostic ECV results in more treatment changes after 3 months, compared to standard of care (no ECV).

Study design: This is an investigator initiated, randomized, open label with blinded endpoint evaluation, multi-centre, trial.

Study population: 112 patients with chronic HF and ECG confirmed persistent AF.

Trial intervention: Patients will be randomized in a 1:1 ratio to either an ECV or standard of care with pharmacological rate and/or rhythm control.

Main study parameters/endpoints:

The primary outcome: total number of treatment alterations by the physician during 3 months post intervention/randomization.

Secondary outcomes: Success rate of ECV, recurrences of AF at 4 weeks, QoL changes assessed by AFEQT and KCCQ score, echocardiographic changes (left ventricular ejection fraction (LVEF) and cardiac output (CO)), and laboratory changes (NT-proBNP) between baseline (pre-cardioversion) and 4 weeks (post-cardioversion). Whether the physician can distinguish AF from HF symptoms and whether ECV can be used as diagnostic tool.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since this is a pragmatic trial, the study will be embedded within care according to current AF and HF guidelines, that includes ECV and rhythm and/or rate control, while acknowledging wide variability in local practises. The patients in the intervention arm will undergo a diagnostic ECV. Both groups will fill out questionnaires regarding QoL (baseline and 4 weeks) and have an echocardiogram at 4 weeks. A blinded endpoint committee will assess potential treatment alterations prescribed by the physician in both patient groups within 3 months. No harm is expected for this study as the intervention will be based on national guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with age ≥ 18 years
2. Diagnosis of HF ≥90 days prior to screening NYHA class ≥ 2 on guideline-directed medical therapy.
3. ECG-confirmed AF/Atrial flutter at screening
4. Received oral anti-coagulants for ≥ 3 weeks (DOAC, vitamin K antagonists with an INR between 2 and 3) prior to screening
5. Patients eligible for both treatment strategies judged by the investigator and physician.
6. Provide written dated informed consent for participation prior to trial admission.

Exclusion Criteria:

A potential patient who meets any of the following criteria will be excluded from participation in this study:

1. Inability to understand and sign informed consent form
2. Hospitalization for acute HF or worsening HF ≤ 3 months prior to screening
3. Heart rate during AF/ atrial flutter ≥ 110 bpm, despite optimal rate control therapy at screening
4. Paroxysmal or permanent AF/atrial flutter
5. Previous left atrial ablation or surgery ≤ 3 months prior to screening
6. Planned catheter ablation at time of screening
7. AF due to a reversible cause (e.g. post-operative AF, hyperthyroidism)
8. Recent acute coronary syndrome, stroke/transient ischemic attack or cardiac intervention (≤90 days). Cardiac interventions include percutaneous coronary intervention, coronary artery bypass grafting, and heart valve repair or replacement (endovascular or surgical)
9. Presence of (or scheduled for) mechanical assist device or heart transplantation
10. Patients with complex congenital heart disease, up to the discretion of the investigator.
11. Patients with current echocardiographic evidence of severe aortic-, mitral-, tricuspid- or pulmonary- valve disease (either stenosis or regurgitation)
12. Patients with an intracardiac thrombus
13. Expected life span from time of enrolment of ≤1 year, as assessed by the clinician
14. Patient currently enrolled in another randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Total number of treatment alterations | During 3 months post intervention/randomization
  Total number of heart failure and/or atrial fibrillation treatment alterations by the physician

SECONDARY OUTCOMES:
Success rate of the ECV | At baseline
  defined as ECG-confirmed sinus rhythm after ECV
Changes in Quality of Life, as assessed by the Atrial Fibrillation Effect on Quality-of-life Questionnaire (AFEQT) questionnaire. | Between baseline and 4 weeks
  Scores range from 0-100. A score of 0 corresponds to complete disability, while a score of 100 corresponds to no disability.
Changes in Quality of Life, as assessed by the The Kansas City Cardiomyopathy Questionnaire (KCCQ) questionnaire | Between baseline and 4 weeks
  Scores range from 0-100, with lower scores corresponding with a poorer Quality of Life. 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Echocardiographic changes, measured by left ventricle ejection fraction (LVEF) | Between baseline and 4 weeks
  Heart failure with reduced ejection fraction (HFrEF); LVEF ≤40%, Heart failure with mid-range ejection fraction (HFmrEF); LVEF 41-49%, Heart failure with preserved ejection fraction (HFpEF); LVEF ≥50%.
Changes in cardiac output, measured using the echocardiographic measurements using velocity time interval. | Between baseline and 4 weeks
Laboratory changes of serum NT pro-BNP levels | Between baseline and 4 weeks
Questioannire physician whether ECV can be used to distinguish AF-specific from HF-specific symptoms | between baseline and 3 months
  10-point likert scale
Time to Photoplethysmography (PPG)-based recurrence of AF (intervention arm). | Between baseline and 3 months
Changes in inflammatory markers | Between baseline and 4 weeks
  To study the association between inflammation and atrial fibrillation, we will measure serum proteins at two different time points, for both the intervention and control group. We will investigate whether inflammatory proteins are different in HF patients who returned to sinus rhythm (the intervention group), compared to patients with persistent atrial fibrillation (standard of care). Moreover, we will asses the effects of electrical cardioversion (intervention group) on plasma proteins over time.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No